CLINICAL TRIAL: NCT00451997
Title: Phase II Trial of Gleevec and Low-Dose Ara-C for Elderly Patients With C-Kit Positive Acute Myeloid Leukemia and High-Risk Myelodysplastic Syndromes
Brief Title: Gleevec/Low-Dose Ara-C Study for Elderly Patients With AML and Myelodysplastic Syndromes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2003-0935
Record Dates: First submitted 2007-03-23; First posted 2007-03-26 (Estimated); Last update posted 2012-08-01 (Estimated); Status verified 2012-07

CONDITIONS: Leukemia, Myeloid; Myelodysplastic Syndromes
Keywords: AML; MDS; Gleevec; Ara-C; C-Kit Positive Acute Myeloid Leukemia; High-Risk Myelodysplastic Syndromes
MeSH Terms: conditions — Leukemia, Myeloid; Myelodysplastic Syndromes | interventions — Imatinib Mesylate; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gleevec + Low-Dose Ara-C (Experimental)
  Interventions: Drug: Gleevec; Drug: Ara-C

INTERVENTIONS:
Drug: Gleevec — 600 mg (capsules) by mouth once daily
  Other Names: Imatinib Mesylate; STI-571; Imatinib; NSC-716051
Drug: Ara-C — 10 mg as an injection under the skin daily for 21 days of every 28 day cycle
  Other Names: Cytarabine; Cytosar-U®; DepoCyt; Cytosine arabinosine hydrochloride; Arabinosylcytosine

SUMMARY:
The goal of this clinical research study is to learn if the combination of Gleevec (imatinib mesylate) and low doses of Cytarabine (ara-C) may help to control leukemia while causing fewer side effects than standard high dose chemotherapy.

DETAILED DESCRIPTION:
Imatinib mesylate is a drug that blocks a certain protein. This protein is thought to be important in the growth of leukemia cells. Ara-C is a chemotherapy drug that has been used for many years to treat AML and MDS.

Imatinib mesylate (Gleevec) is a protein-tyrosine kinase inhibitor that inhibits the Bcr-Abl tyrosine kinase, as well as the receptor tyrosine kinases for platelet- derived growth factor (PDGF) and stem cell factor (SCF), c-Kit, and inhibits PDGF- and SCF-mediated cellular events. c-Kit is expressed in over 90% of patients with AML.

The treatment of AML for patients age 65 or older with AML or high-risk MDS (age ³ 60 if high-risk cytogenetics) have a poor prognosis with induction chemotherapy. Response rate is no more than 45% with an induction mortality of at least 25%, and 1-year survival no better than 20%. Indeed, most patients in these age groups are not even offered therapy and are managed with supportive care only. Thus, new therapies that are better tolerated are needed.

Imatinib alone can induce response in nearly 20% of patients, and there is synergy with low concentrations of ara-C. In this study we plan to investigate the combination of imatinib and low-dose ara-C.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are not candidates for intensive chemotherapy with any of the following diagnosis: 1. AML or MDS (with >/=5% blasts) age >/= 65 years old (or age >/= 60 if high-risk cytogenetics), or 2. AML or MDS (RAEB or RAEBT) of any cytogenetic group age 60 or older with minimally treated disease who have relapsed disease or are refractory to therapy and not likely to require cytoreductive therapy within one month, and, or 3. CMML.
* Patients with WHO performance status of 0 to 2
* Patients must have recovered from prior cytotoxic chemotherapy; treatment with hydrea is allowed up to 24 hours prior to day 1 of study drug administration
* Written informed consent obtained according to local guidelines
* Patients must have a serum creatinine of </= 1.5 x ULN, SGPT </= 3 x ULN and total bilirubin </= 2.0 x ULN.
* Patients with >/= 20% blasts positive for c-kit (CD117) (except for CMML)
* Postmenopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential. Male and female patients of childbearing potential must agree to employ an effective method of birth control throughout the study and for up to 3 months following discontinuation of study drug.

Exclusion Criteria:

* Patients with uncontrolled active infection
* Patients with NYHA class III or IV
* Women who are pregnant
* Women who are breast feeding

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2004-03; Primary Completion 2005-08 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Efficacy of a combination of imatinib and low dose ara-C in elderly or high-risk patients with AML and MDS, as measured by the rate of early mortality or progression. | April 2007

SECONDARY OUTCOMES:
Rate of overall response, including CRp and PR. | April 2007
To determine the safety profile of this combination. | April 2007
To determine the impact on long-term survival of this therapy. | April 2007
To determine the duration of responses obtained with this therapy. | April 2007
To determine the impact of this therapy in cognitive function. | April 2007
To determine the effect of this approach in quality of life of this patient population. | April 2007
To determine the overall costs (health economic analysis) associated with this combination therapy. | April 2007

CONTACTS AND LOCATIONS:
Overall Officials: Jorge E Cortes, MD, Principal Investigator — The University of M.D. Anderson Cancer Center
Locations (1):
- The University of Texas M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M.D. Anderson's website — http://mdanderson.org